CLINICAL TRIAL: NCT06447792
Title: Survival Rate of 2 Implant-supported Short-span Fixed Partial Dentures in the Anterior Mandible: A Retrospective Study
Brief Title: Survival Rate of 2 Implant-supported Short-span Fixed Partial Dentures
Status: Recruiting | Type: Observational
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Mohammed El-Sawy, lecturer, Department of Prosthodontics, principle investigator, Menoufia University
Other Study IDs: ADMNF-0020524
Record Dates: First submitted 2024-06-02; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Implant Complication; Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: immediately placed implants with a delayed loading protocol. Loading was performed after 3 months.
  Interventions: Other: Loading protocol
- Group 2: immediately placed implants with a progressive loading protocol. Loading was performed after 5 weeks.
  Interventions: Other: Loading protocol
- Group 3: immediately placed implants with an immediate loading protocol. The day of the surgery was also the day of loading.
  Interventions: Other: Loading protocol

INTERVENTIONS:
Other: Loading protocol — The prosthetic restoration and functional loading of the dental implant.

SUMMARY:
Implant supported superstructure is necessary for long term success and durability of the implant itself in terms of stresses distribution and fracture strength capability.1 Stresses falling on an implant are too much greater than those applied on a tooth structure with a periodontal ligament offering a degree of elasticity. The important mechanical and physical properties of materials used for the fabrication of dental prostheses include adequate flexural and tensile strength and modulus of elasticity, maximum fracture resistance, optimal bond strength and adequate polishability.

DETAILED DESCRIPTION:
The relationship between implants/ prosthetic components and the surrounding soft and hard tissues is complex and determines the final clinical result. For example, crestal bone resorption, frequently observed following implant placement or following loading, may be related to factors such as the establishment of the biologic width, the macro design of the cervical area of the implant and possible surface treatments, the type of implant/abutment connection, the positioning of the implant in relation to the bone crest, the width of the alveolar ridge, the distance between contiguous implants, the surgical procedure, and the effects of overloading and peri-implantitis. The establishment of the biologic width perse is related to a series of events that results in remodeling of the bone that surrounds the implants, a fact that has been observed by histomorphometry and radiographic analysis.

The aim of the present study was to compare and evaluate the survival rate and crestal bone levels around immediately placed implants in the esthetic zone with delayed, progressive, or immediately placed.

ELIGIBILITY:
Inclusion Criteria:

* fully dentulous people over 25 who complained of the mobility of 4 mandibular incisor teeth, or partially dentulous people who missed 2 mandibular central incisor teeth and had periodontally affected the neighboring lateral incisor teeth.
* These individuals were subsequently treated with 2 implants supporting FPDs and following a delayed, progressive, or immediate loading protocol
* Class 0 or 1 bone defects after tooth extraction, were only included in the study
* The medical records included data regarding implant type, width, and length, surgical procedure, annual hygienist treatments, radiographs, and implant insertion date

Exclusion Criteria:

* had less than 1 years of follow-up, had incomplete restorative or surgical data, had non-diagnostic radiographs, had more or less than 4 unit fixed partial denture
* patients did not present for annual follow-up visits to evaluate oral hygiene measures or treat mechanical or technical complications.
* Individuals with bone defects class 2, 3, 4, or 5 after mandibular lateral incisor tooth extraction were also excluded.

Ages: 25 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People over 25 and less than 50 years
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-08-04 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Implant survival | 3 years
  The implant is present at the follow-up examination but its condition is not specified.

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammed A. Elsawy, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No
For a reasonable reason after contacting the corresponding author.